CLINICAL TRIAL: NCT07097116
Title: The Effect of Structured Exercises Applied in Addition to Hiking Bench Exercise Training on Hiking Endurance and Muscle Activation in Young Sailors
Brief Title: The Effect of Two Different Exercise Programs in Young Sailors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IstinyeU-HPekeren-001
Record Dates: First submitted 2025-07-21; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Healty Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hiking Bench Exercises (Active Comparator): Hiking Bench Training Only Participants will receive an 8-week hiking bench training program, based on Laser Pro Hikingbench™ exercises. The protocol includes progressive static, dynamic endurance and strength tasks mimicking hiking postures in sailing.
  Interventions: Other: Hiking Bench Exercise Program
- Hiking Bench + Structured Exercise Program (Experimental): Participants will receive the same 8-week hiking bench protocol as Arm 1, plus an additional structured exercise program targeting aerobic capacity, core stability, balance, and motor competence.
  Interventions: Other: Structured Land-Based Exercise Program

INTERVENTIONS:
Other: Hiking Bench Exercise Program — The training is performed 2 times per week over 8 weeks. It includes 4 progressive phases using a hiking bench, simulating hiking posture exercises targeting endurance, trunk control, and leg strength.
  Arms: Hiking Bench Exercises
Other: Structured Land-Based Exercise Program — This protocol adds aerobic warm-up, dynamic stretching, foundational strength (glutes, core), and cool-down flexibility work. Exercises are adapted to sailing-specific demands and performed 2 times per week alongside hiking bench work.
  Arms: Hiking Bench + Structured Exercise Program

SUMMARY:
This study aims to investigate the effects of an 8-week structured land-based exercise program on hiking endurance, core endurance, muscle activation, balance, and motor competence in young sailors. The intervention will be applied in addition to a standard hiking bench training, which simulates the physically demanding "hiking" maneuver used in sailing. A total of 26 adolescent athletes, aged 12 to 18 years, will be randomly assigned to two groups: one receiving hiking bench training only, and the other receiving hiking bench training combined with structured strength, flexibility, balance, and dynamic warm-up exercises. Evaluations will include endurance testings, electromyography (EMG) analysis of muscle activity, balance tests, and motor coordination assessments. The results are expected to inform future training programs by optimizing athletic performance and supporting injury prevention strategies in youth sailing.

ELIGIBILITY:
Inclusion Criteria:

* Being between 12 and 18 years old
* Having been involved in sailing for at least 2 years
* Competing at the national or international level
* Being in a sailing class that uses trapeze maneuvers

Exclusion Criteria:

* Having had any upper or lower extremity injury in the last 8 weeks
* Having had any upper or lower extremity surgery in the last 6 months
* Having received land-based exercise training in sailing in the last 4 weeks.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Hiking endurance with incremental resistance | pre-treatment (week 0) and after-treatment (week 8)
  This test is a maximal incremental trapezius endurance test based on the protocol developed by Tan and colleagues. Each participant will sit on a raised, padded bench with their knees extended and the backs of their knees touching the edge of the bench. Instead of a bar, a steel bucket equipped with a padded strap (total weight 1.4 kg) will be attached to the participant's ankles. Since the test is conducted with young sailors, the starting load will be reduced from 15 kg to 0 kg. Participants will maintain a knee angle greater than 130° (monitored throughout the test using an electrogoniometer), and 5 kg plates will be added to the bucket every minute until the subject can no longer hold the weight at the prescribed angle. Participants will be allowed to support themselves by gripping the bench or shifting the load from one leg to the other. They will be verbally encouraged throughout the test. Final endurance times will be recorded in seconds. (Bahchevanski, 2017; Callewaert et al.,

SECONDARY OUTCOMES:
Muscle Activation Measurement | Time Frame: pre-treatment (week 0) and Post-treatment (week 8)
  Muscle activation will be measured using the Noraxon Ultium EMG system. Data will be collected at 1500 Hz using 2.0 cm spaced surface electrodes placed bilaterally on rectus abdominis, rectus femoris, and vastus lateralis muscles. Skin will be shaved, abraded, and cleaned to keep impedance below 5 kΩ. Participants will perform four 3-minute trapeze holds with 15-second rest intervals. During the test, they will extend hip and knee joints to maintain angles of at least 120° and 140°, respectively, while keeping arms crossed over the chest. Raw EMG signals will be band-pass filtered (10-500 Hz), and RMS values will be calculated with a 50 ms sliding window. Signals will be normalized to %MVC using isometric contraction tests. Fatigue will be evaluated by analyzing the slope of RMS over time and by tracking changes in median and mean frequencies using Fast Fourier Transform.
McGill Core Endurance Tests | pre-treatment (week 0 ) and post Treatment (week8)
  McGill's tests will assess core endurance using four positions: trunk flexor, right and left side plank, and trunk extensor. Each participant performs a brief practice, then holds each static position as long as possible. Time is recorded with a stopwatch using "start" and "stop" commands. Test order is randomized. In the flexor test, participants sit with trunk at 60°, knees at 90°, arms crossed; time stops if angle is lost. In side planks, feet are stacked, bottom elbow on the mat, top hand on opposite shoulder; time ends when body alignment is lost. In the extensor test, participants lie prone on a table with ASIS at the edge, arms resting forward. Lower limbs are stabilized with straps or by an assistant. Time starts when arms cross over the chest and trunk is held horizontal, and stops when the posture can't be maintained.
Balance Assessment | pre-treatment (week 0 ) and post-treatment (week 8)
  The modified Y-Balance Test (mYBT) will be used to assess dynamic balance of both legs. Three marked measuring tapes will be placed from the center of the foot in anterior (ANT, 90°), posterolateral (PL, 45°), and posteromedial (PM, 45°) directions. Participants will stand on one leg with a semi-flexed knee and hands on hips, and reach as far as possible in each direction with the other leg. They will lightly touch the furthest point with minimal pressure using the farthest part of the reaching foot, without using it for support. After a 5-minute familiarization, three trials per direction will be performed. The maximum reach in each direction will be recorded. This value will be divided by leg length and multiplied by 100 to calculate relative reach distance.
Motor Competence Assessment | pre-treatment (week0) and post-treatmen (week 8)
  Gross motor coordination will be assessed using the KTK3+ test, which includes three tasks:
  Jumping Sideways (JS): Participants jump sideways over a wooden slat with both feet for 15 seconds. The total score is the sum of jumps from two trials.
  Moving Sideways (MS): Participants move laterally by stepping on and shifting two wooden boards for 20 seconds. The score is the total number of board shifts and steps from two trials.
  Balancing Backwards (BB): Participants walk backward on three beams of decreasing width (6.0 cm, 4.5 cm, 3.0 cm). Three trials per beam are performed. The maximum score is 72 steps.
  Eye-Hand Coordination (EHC): In a 30-second task, participants throw a tennis ball with one hand and catch it with the other, alternating hands. Standing 1 meter from a 1 m² wall square, they perform two trials. Total successful catches are recorded as the score.

CONTACTS AND LOCATIONS:
Overall Officials: Berrak Varhan, Study Chair — Istinye University

IPD SHARING:
Plan to Share IPD: Yes
The study will share de-identified, summary-level outcome data, including group-level means, standard deviations, effect sizes, and p-values derived from statistical analyses. These data will be provided to support transparency and allow for interpretation of the study findings.
Supporting Information: Study Protocol, SAP
Time Frame: Summary-level data and supporting documents (e.g., study protocol and statistical analysis plan) will be available within 12 months following the final publication of study results and will remain accessible for at least 5 years via institutional repository or upon reasonable request.
Access Criteria: The study's outcome results, including group-level means, standard deviations, p-values, and effect sizes, as well as supporting materials such as the study protocol and statistical analysis plan, will be made available to qualified academic researchers upon reasonable request. Data will be provided for ethically approved, non-commercial research purposes. Interested investigators should contact the principal investigator through the affiliated institution and submit a written request describing the intended use and data handling procedures. Each request will be reviewed individually in accordance with institutional data-sharing guideline.

REFERENCES:
- [Background] Tan B, Aziz AR, Spurway NC, Toh C, Mackie H, Xie W, Wong J, Fuss FK, Teh KC. Indicators of maximal hiking performance in Laser sailors. Eur J Appl Physiol. 2006 Sep;98(2):169-76. doi: 10.1007/s00421-006-0260-3. Epub 2006 Aug 3. PMID 16896729
- [Background] Callewaert M, Boone J, Celie B, De Clercq D, Bourgois JG. Indicators of sailing performance in youth dinghy sailing. Eur J Sport Sci. 2015;15(3):213-9. doi: 10.1080/17461391.2014.905984. Epub 2014 Apr 10. PMID 24720497
- [Background] Pan D, Sun K, Liu X. Adjunctive hiking bouts during 8 weeks regular sailing training improves cardiorespiratory and muscular responses during hiking emulation in highly trained sailors. Eur J Sport Sci. 2024 Jul;24(7):878-888. doi: 10.1002/ejsc.12118. Epub 2024 May 17. PMID 38956795
- See also: Source of protocol of Bucket test — https://www.researchgate.net/publication/340903820_DETERMINATION_THE_MAIN_INDICATORS_OF_SAILING_PERFORMANCE_IN_OPTIMIST_SAILOR'S